CLINICAL TRIAL: NCT01192568
Title: A Two-part, Multicenter, Dose-titration Study Evaluating the Efficacy, Safety, Pharmacodynamics and Pharmacokinetics of Oxybutynin Chloride 10% Gel for the Treatment of Detrusor Overactivity Associated With a Neurological Condition in Pediatric Patients
Brief Title: Safety and Efficacy Evaluation of Oxybutynin Topical Gel In Children With Neurogenic Bladder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OG09002
Record Dates: First submitted 2010-08-30; First posted 2010-09-01 (Estimated); Results first posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Overactive Detrusor; Neurogenic Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Bladder, Neurogenic | interventions — oxybutynin

STUDY DESIGN:
Intervention Model Description: This study was initiated as a double-blind, placebo-controlled study with an open-label extension and was amended (in Protocol Amendment 3) to continue to enroll subjects under only open-label treatment.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Pre-Amendment 3: All subjects, site personnel and Watson and CRO personnel directly involved in the execution of the study were blinded. Post-Amendment 3: All subjects Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- DB: OTG (Pre-Amend 3) (Experimental): Double-Blind Oxybutynin Chloride topical gel (OTG) (Pre-Amendment 3) Oxybutynin Chloride topical gel (OTG), 0.5 g, 0.75 g (starting dose), or 1 g sachets, applied transdermally once daily for 6 weeks.
  Followed by OL OTG for 8 weeks.
  Interventions: Drug: Oxybutynin
- OL: OTG (Post-Amend 3) (Experimental): Open-Label Oxybutynin Chloride topical gel (OTG) (Pre & Post-Amendment 3) Oxybutynin Chloride topical gel (OTG), 0.5 g, 0.75 g (starting dose for Pre- and Post-Amendment 3), or 1 g sachets, applied transdermally once daily for 14 weeks.
  Interventions: Drug: Oxybutynin
- DB: Placebo (Pre-Amend 3) (Placebo Comparator): Double-Blind Placebo (Pre-Amendment 3) Placebo Gel sachets applied transdermally once daily for 6 weeks. Followed by OL OTG for 8 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxybutynin — 10% Oxybutynin Chloride Topical Gel, 0.5 g, 0.75 g, and 1 g/day, administered transdermally.
  Other Names: Gelnique
  Arms: DB: OTG (Pre-Amend 3); OL: OTG (Post-Amend 3)
Drug: Placebo — Topical gel
  Arms: DB: Placebo (Pre-Amend 3)

SUMMARY:
This study will evaluate the safety and efficacy of Oxybutynin Chloride 10% Topical Gel in children 3 to less than 17 years old, who have overactive bladder due to a neurogenic condition. Children will be treated with 0.75 g of gel/day for two weeks. Patients will then return to the clinic for a potential dose titration. At this time their dose may be adjusted up to 1g/day, down to 0.5g/day, or remain the same at 0.75g of gel/day depending on the individual response and tolerability. The total treatment time is 14 weeks and total time on the study is 16 weeks.

DETAILED DESCRIPTION:
This study will use a two-part, multicenter, dose-titration study in pediatric patients with a detrusor overactivity associated with a neurological condition

ELIGIBILITY:
Inclusion Criteria:

* 3 years to < 17 years
* Neurogenic bladder
* Neurological condition
* CIC

Exclusion Criteria:

* Have anatomical bladder abnormalities
* Sensitivity to anticholinergics
* Bladder augmentation

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2011-05-17 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2023-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (10):
- United States (10):
  - Loma Linda University /ID# 236889, Loma Linda, California
  - Child Hosp of Orange County,CA /ID# 237517, Orange, California
  - Children's Hospital Colorado - Aurora /ID# 237620, Aurora, Colorado
  - Augusta University Medical Center /ID# 238188, Augusta, Georgia
  - University of Mississippi Medical Center /ID# 238065, Jackson, Mississippi
  - Albany Medical College /ID# 236880, Albany, New York
  - Duke University /ID# 237494, Durham, North Carolina
  - Duplicate_Oregon Health & Science University /ID# 234354, Portland, Oregon
  - Cook Children's Med. Center /ID# 237538, Fort Worth, Texas
  - Child Hosp of the King's Dtr's /ID# 237799, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Background] Cartwright PC, Coplen DE, Kogan BA, Volinn W, Finan E, Hoel G. Efficacy and safety of transdermal and oral oxybutynin in children with neurogenic detrusor overactivity. J Urol. 2009 Oct;182(4):1548-54. doi: 10.1016/j.juro.2009.06.058. Epub 2009 Aug 15. PMID 19683731

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This 2-part pediatric study, was initiated as a double-blind (DB), placebo-controlled study with an open-label (OL) extension (Protocol Amendment 3). In Part 1 (Pre-Amendment 3), subjects were randomized into DB: Placebo (Pre-Amend 3) or DB: OTG (Pre-Amend 3) treatment groups for 6 weeks, then all subjects were placed into OL: OTG (Pre-Amend 3) for 8 weeks. In Part 2 (Post-Amendment 3), newly enrolled subjects were placed into OL: OTG (Post-Amend 3) for 14 weeks.
Groups:
- DB: Placebo (Pre-Amend 3): Subjects were randomized to receive Double-Blind (DB) placebo gel for 6 weeks.
  Followed by:
  OL oxybutynin chloride gel (OTG) for 8-week period to generate additional safety data.
- DB: OTG (Pre-Amend 3): Subjects were randomized to receive DB oxybutynin chloride gel (OTG) for 6 weeks.
  All subjects began treatment with 0.75 g of gel/day for 2 weeks. The dose of OTG was adjusted to obtain the optimal clinical response. The dose titration of OTG could be adjusted up to 1 g/day, down to 0.5 g/day, or remain the same at 0.75 g/day.
  Followed by:
  OL OTG for 8-week period to generate additional safety data.
- OL: OTG (Pre-Amend 3): Following the DB Period:
  Subjects received Open-Label (OL) oxybutynin chloride gel (OTG) for 8 weeks.
  All subjects began treatment with 0.75 g of gel/day for 2 weeks. The dose of OTG was adjusted to obtain the optimal clinical response. The dose titration of OTG could be adjusted up to 1 g/day, down to 0.5 g/day, or remain the same at 0.75 g/day.
- OL: OTG (Post-Amend 3): Subjects received OL oxybutynin chloride gel (OTG) for 14 weeks.
  All subjects began treatment with 0.75 g of gel/day for 2 weeks. The dose of OTG was adjusted to obtain the optimal clinical response. The dose titration of OTG could be adjusted up to 1 g/day, down to 0.5 g/day, or remain the same at 0.75 g/day.
Period: Double Blind Pre-Amendment 3
Arm/Group | DB: Placebo (Pre-Amend 3) | DB: OTG (Pre-Amend 3) | OL: OTG (Pre-Amend 3) | OL: OTG (Post-Amend 3)
Started | 16 | 17 | 0 | 0
Completed | 16 | 17 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Open Label Pre-Amendment 3
Arm/Group | DB: Placebo (Pre-Amend 3) | DB: OTG (Pre-Amend 3) | OL: OTG (Pre-Amend 3) | OL: OTG (Post-Amend 3)
Started | 0 | 0 | 33 | 0
Completed | 0 | 0 | 32 | 0
Not Completed | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0
Period: Open Label Post-Amendment 3
Arm/Group | DB: Placebo (Pre-Amend 3) | DB: OTG (Pre-Amend 3) | OL: OTG (Pre-Amend 3) | OL: OTG (Post-Amend 3)
Started | 0 | 0 | 0 | 19
Completed | 0 | 0 | 0 | 18
Not Completed | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DB: Placebo (Pre-Amend 3) | DB: OTG (Pre-Amend 3) | OL: OTG (Post-Amend 3) | Total
Number analyzed (Participants) | 16 | 17 | 19 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.7 (3.11) | 9.6 (2.71) | 7.7 (3.41) | 9.0 (3.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 10 | 28
  Male | 8 | 7 | 9 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 7 | 16
  Not Hispanic or Latino | 11 | 13 | 12 | 36
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 4 | 5 | 1 | 10
  White | 10 | 11 | 15 | 36
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 1 | 0 | 0 | 1
Percent of Catheterizations without Leaking Week 0 (Baseline) [Mean (Standard Deviation); unit: percentage of catheterizations wo leak] — Population: ITT Population
  percentage of catheterizations wo leak
    number analyzed (Participants) | 16 | 17 | 18 | 51
    (all) | 32.98 (32.708) | 27.88 (35.225) | 18.63 (27.078) | 23.12 (31.185)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Percent of Catheterizations Without a Leaking Accident at Week 6
Description: The primary efficacy endpoint is the change from baseline to Week 6 of treatment or the last observation carried forward in percentage of catheterizations without a leaking accident as recorded in a 2-day urinary diary.
Time Frame: Baseline (Week 0) up to Week 6
Population: ITT Population
Measure: Mean (Standard Deviation); unit: percentage of point
Groups:
- Placebo: Subjects were randomized to receive Double-Blind (DB) placebo gel for 6 weeks.
  Followed by:
  OL oxybutynin chloride gel (OTG) for 8-week period.
- OTG (Pre-Amend 3): All randomized subjects who have at least 1 post-baseline value for efficacy variable for both the DB and OL periods before Protocol Amendment 3.
  Subjects were randomized to receive DB oxybutynin chloride gel (OTG) for 6 weeks.
  All subjects began treatment with 0.75 g of gel/day for 2 weeks. The dose of OTG was adjusted to obtain the optimal clinical response. The dose titration of OTG could be adjusted up to 1 g/day, down to 0.5 g/day, or remain the same at 0.75 g/day.
  Followed by:
  OL OG for 8-week period.
- OTG (Post-Amend 3): All subjects who receive at least 1 dose of study treatment and have at least 1 post-baseline value for the efficacy variable in the Post-Amendment 3 OL period. Subjects received OL oxybutynin chloride gel (OTG) for 14 weeks. All subjects began treatment with 0.75 g of gel/day for 2 weeks. The dose of OTG was adjusted to obtain the optimal clinical response. The dose titration of OTG could be adjusted up to 1 g/day, down to 0.5 g/day, or remain the same at 0.75 g/day.
- Combined OTG: All subjects who receive at least 1 dose of study treatment and have at least 1 post-baseline value for the primary efficacy variable in the Post-Amendment 3 open-label period and all randomized subjects who have at least 1 post-baseline value for the efficacy variable in the Pre-Amendment 3 double-blind period.
Arm/Group | Placebo | OTG (Pre-Amend 3) | OTG (Post-Amend 3) | Combined OTG
Number analyzed (Participants) | 16 | 17 | 18 | 35
percentage of point | -0.45 (20.178) | 16.91 (36.681) | 13.82 (22.978) | 15.32 (29.994)
Statistical Analysis 1: Comparison: Placebo vs Combined OTG; Test type: Superiority; p = 0.0928, ANCOVA; Mean Difference (Final Values) = 14.22, 95% CI 2-sided [-2.45 to 30.90], Standard Error of Mean 4.612

2. Secondary Outcome: Change From Baseline in Average Volume of Urine Collected Per Catheterization at Week 6
Description: Pre-Amendment 3:
  Change from Baseline in Average Volume of Urine Collected per Catheterization at week 6 (calculated from the 2-day urinary diary data).
Time Frame: Baseline (Week 0) up to week 6
Population: ITT Population
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Placebo | OTG (Pre-Amend 3)
Number analyzed (Participants) | 16 | 17
mL | -24.59 (38.138) | 14.33 (38.781)
Statistical Analysis 1: Comparison: OTG (Pre-Amend 3); Test type: Superiority; p = 0.0054, ANCOVA; Mean Difference (Final Values) = 34.92, 95% CI 2-sided [11.13 to 58.70], Standard Error of Mean 8.089

3. Secondary Outcome: Change From Baseline in Average Volume of Urine Collected Per First (Morning Awakening) Catheterization at Week 6
Description: Change from Baseline in Average Volume of Urine Collected Per First (Morning Awakening) Catheterization at week 6 (calculated from the 2-day urinary diary data).
Time Frame: Baseline (Week 0) up to Week 6
Population: ITT Population
Measure: Mean (Standard Deviation); unit: mL
Groups:
- OTG (Pre-Amend 3): All randomized subjects who have at least 1 post-baseline value for efficacy variable for both the DB and OL periods before Protocol Amendment 3. Subjects were randomized to receive DB oxybutynin chloride gel (OTG) for 6 weeks.
  All subjects began treatment with 0.75 g of gel/day for 2 weeks. The dose of OTG was adjusted to obtain the optimal clinical response. The dose titration of OTG could be adjusted up to 1 g/day, down to 0.5 g/day, or remain the same at 0.75 g/day.
  Followed by:
  OL OTG for 8-week period.
Arm/Group | Placebo | OTG (Pre-Amend 3) | OTG (Post-Amend 3) | Combined OTG
Number analyzed (Participants) | 16 | 17 | 18 | 35
mL | -12.03 (88.116) | 14.18 (58.694) | 29.78 (87.808) | 22.20 (74.424)
Statistical Analysis 1: Comparison: Combined OTG; Test type: Superiority; p = 0.1739, ANCOVA; Mean Difference (Final Values) = 32.59, 95% CI 2-sided [-14.89 to 80.07], Standard Error of Mean 13.215

4. Secondary Outcome: Change From Baseline in Average Number of Catheterizations Per Day at Week 6
Description: Change from Baseline in Average Number of Catheterizations Per Day at Week 6 (calculated from the 2-day urinary diary data).
Time Frame: Baseline (Week 0) up to Week 6
Population: ITT
Measure: Mean (Standard Error); unit: Number of Catheterizations Per Day
Groups:
- Combine OTG: All subjects who receive at least 1 dose of study treatment and have at least 1 post-baseline value for the primary efficacy variable in the Post-Amendment 3 open-label period and all randomized subjects who have at least 1 post-baseline value for the efficacy variable in the Pre-Amendment 3 double-blind period.
Arm/Group | Placebo | OTG (Pre-Amend 3) | OTG (Post-Amend 3) | Combine OTG
Number analyzed (Participants) | 16 | 17 | 18 | 35
Number of Catheterizations Per Day | 0.19 (0.512) | -0.03 (0.450) | -0.67 (0.924) | -0.36 (0.791)
Statistical Analysis 1: Comparison: OTG (Pre-Amend 3); Results from a pre-specified test (Kolmogorov-Smirnov test p <= 0.05) determined that the Pre-Am3 and Post-Am3 OTG data should be analyzed separately for the primary analysis; Test type: Superiority; p = 0.2660, ANCOVA; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.53 to 0.15], Standard Error of Mean 0.117
Statistical Analysis 2: Comparison: OTG (Post-Amend 3); Test type: Superiority; p = 0.0070, t-test, 2 sided; Mean Difference (Final Values) = -0.67, 95% CI 2-sided [-1.13 to -0.21]

ADVERSE EVENTS:
Time Frame: All-cause mortality were reported from enrollment to the end of study, median time on follow up was 42.0,43.0, 57.0, and 99.0 days for DB: Placebo (Pre-Amend 3), DB: OTG (Pre-Amend 3) OL: OTG (Pre-Amend 3), and OL: OTG (Post-Amend 3), respectively.
Description: Treatment-emergent adverse events and serious adverse events were collected from first dose of study drug until 2 weeks after the last dose of study drug; mean duration on study drug was 42.1, 56.0, and 96.6 days for DB: Placebo (Pre-Amend 3), OTG (Pre-Amend 3), and OL: OTG (Post-Amend 3) , respectively.
Groups:
- DB: OTG (Pre-Amend 3): Subjects were randomized to receive DB oxybutynin chloride gel (OTG) for 6 weeks.
  All subjects began treatment with 0.75 g of gel/day for 2 weeks. The dose of OTG was adjusted to obtain the optimal clinical response. The dose titration of OTG could be adjusted up to 1 g/day, down to 0.5 g/day, or remain the same at 0.75 g/day.
  Followed by:
  OL OG for 8-week period to generate additional safety data.
- OL: OTG (Pre-Amend 3): Subjects received Open-Label (OL) oxybutynin chloride gel (OTG) for 8 weeks.
  All subjects began treatment with 0.75 g of gel/day for 2 weeks. The dose of OTG was adjusted to obtain the optimal clinical response. The dose titration of OTG could be adjusted up to 1 g/day, down to 0.5 g/day, or remain the same at 0.75 g/day.
Arm/Group | DB: Placebo (Pre-Amend 3) | DB: OTG (Pre-Amend 3) | OL: OTG (Pre-Amend 3) | OL: OTG (Post-Amend 3)
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/17 | 0/33 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/17 | 3/33 | 3/19
Other Adverse Events (participants affected / at risk) | 8/16 | 12/17 | 16/33 | 15/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DB: Placebo (Pre-Amend 3) (N=16) | DB: OTG (Pre-Amend 3) (N=17) | OL: OTG (Pre-Amend 3) (N=33) | OL: OTG (Post-Amend 3) (N=19)
INGUINAL HERNIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
UROSEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LIMB DEFORMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DEVICE MALFUNCTION (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DB: Placebo (Pre-Amend 3) (N=16) | DB: OTG (Pre-Amend 3) (N=17) | OL: OTG (Pre-Amend 3) (N=33) | OL: OTG (Post-Amend 3) (N=19)
TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DRY EYE (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OPTIC DISC DRUSEN (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VISION BLURRED (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
ANAL INCONTINENCE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DRY MOUTH (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
VOMITING (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
ASTHENIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FEELING HOT (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
ASYMPTOMATIC BACTERIURIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CELLULITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CONJUNCTIVITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
EAR INFECTION (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
GASTROENTERITIS VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INFLUENZA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ORAL HERPES (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTITIS MEDIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PHARYNGITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SINUSITIS (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 3 (3) | 2 (2) | 4 (4) | 4 (4)
URINARY TRACT INFECTION ENTEROCOCCAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VIRAL PHARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CONTUSION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LIMB INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SCRATCH (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SKIN WOUND (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BLOOD POTASSIUM INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NEUTROPHIL COUNT INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
JOINT CONTRACTURE (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
JOINT EFFUSION (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
TENDINOUS CONTRACTURE (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
ANXIETY (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ATTENTION DEFICIT HYPERACTIVITY DISORDER (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INSOMNIA (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BLADDER DISCOMFORT (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MICTURITION URGENCY (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
URINE ABNORMALITY (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GENITAL RASH (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VULVOVAGINAL ERYTHEMA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ECZEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SKIN EXFOLIATION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
COLOSTOMY (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FLUSHING (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
HYPERTENSION (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
AbbVie has decided to discontinue further subject enrollment in the OG09002 (Oxybutynin) study. This decision is not based on a safety or an efficacy signal; rather this decision was made because of a change in AbbVie's development.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-10-31): https://cdn.clinicaltrials.gov/large-docs/68/NCT01192568/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-28): https://cdn.clinicaltrials.gov/large-docs/68/NCT01192568/SAP_001.pdf